CLINICAL TRIAL: NCT02291146
Title: LA Sprouts: The Impact of Gardening and Nutrition Education on Childhood Obesity in Latino Youth
Acronym: LA Sprouts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Loma Linda University (Other); University of Texas at Austin (Other); University of California, Los Angeles (Other); National Institutes of Health (NIH) (NIH); Annenberg Foundation (Unknown)
Responsible Party: Principal Investigator, Donna Spruijt-Metz, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIH R21 DK094066-02
Record Dates: First submitted 2014-10-24; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Pediatric Obesity
Keywords: gardening; cooking; nutrition education; Hispanic Americans
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LA Sprouts intervention (Experimental): The intervention classes will be taught during a 90-minute session once a week for 12 weeks. Participants will receive a 45-minute gardening lesson, taught by a Master Gardener (supervised by Dr. Gatto). This lesson will include learning how to plant, maintain and harvest various fruits and vegetables. Supplementing the gardening lesson, a USC nutrition educator, with help from various graduate students (supervised by PI Dr. Davis), will lead a 45-minute cooking activity and nutrition education lesson. Every participant will participate in the cooking activity and sample the food. The program will include lessons on growing crops that have cultural significance to Latino youth such as nopales, beans, corn and squash (the latter three crops are commonly referred to as "the three sisters").
  Interventions: Behavioral: LA Sprouts intervention
- control (No Intervention): Approximately 200 students in the second region who are enrolled in LA's Best will serve as control participants. After the 12-week intervention is conducted and all post-testing measures are collected on controls, a vegetable/fruit garden will be built at both control schools and the LA Sprouts program will be taught to all 3rd, 4th and 5th graders in LAs Best and their parents at the control school as a delayed intervention.

INTERVENTIONS:
Behavioral: LA Sprouts intervention — see arm 1 description
  Arms: LA Sprouts intervention

SUMMARY:
The overall goal of this project is to conduct a randomized controlled 12-week after school, gardening, nutrition and cooking program (called "LA Sprouts") to improve dietary intake and reduce obesity in 3rd, 4th and 5th grade students (ages 8-12 years) in Los Angeles. Approximately 400 3rd - 5th grade students participating in the LA's Best after school program will participate. Four elementary schools in Los Angeles will be selected to participate in the study. Schools will be randomized by region to either receive the intervention (LA Sprouts; 2 schools, n=200 students) or serve as controls (received a delayed intervention program one school semester later; 2 schools, n=200 students). The LA Sprouts intervention will take place at the elementary schools, with gardens on campus specially designed and built for this project. The program will be held once a week for 12 weeks and will consist of a 45-minute gardening lesson, taught by Master Gardeners from the University of California Cooperative Extension (supervised by Nicole Gatto, MPH, PhD), and a 45-minute nutrition education and cooking lesson, taught by USC a Nutrition Educator (supervised by Jaimie Davis, PhD, RD). Measures of childhood obesity (i.e., body mass index (BMI) and body fat percentages), blood pressure, metabolic function (fasting blood glucose, insulin and lipids), dietary intake and related behaviors, and school performance will be measured before and after the implementation of the program in both intervention and control participants. Approximately 10 additional students of the same age will be asked to participate in a focus group to evaluate the questionnaire developed for this study. In addition, approximately 20 additonal students of the same age will be asked to participate in a test-retest session to validate the reliability of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Normal, Overweight and Obese Children: Investigators will attempt to obtain a natural selection of normal weight children (age- & sex-specific BMI < 85th percentile based on CDC BMI growth charts (40) and overweight and obese children (BMI ≥ 85th percentile). Based on preliminary data from these areas, investigators expect that at least 50% of the sample will be overweight or obese. There will not be an upper BMI limit.

Gender & Age: Investigators will attempt to enroll equal numbers of female and male students in 3rd through 5th grades (8-12 years of age).

Latino origin: This study will include all ethnicities, however the selected schools are >90% Latino.

Exclusion Criteria:

* The following criteria are exclusionary: presently taking medication(s) or diagnosed with any disease that could influence dietary intake or body composition; previously diagnosed with any major illness since birth (e.g. chronic birth asphyxia, cancer, etc.); any physical, cognitive, or psychological disability that would prevent participation in the study. Participants testing positive for diabetes (as determined from the fasting blood draw) will be referred for treatment. (Note: subjects with pre-diabetes will be eligible for the study). Although participant data may be excluded based on the above exclusion criteria, participation in the program classes may be allowed. Individual cases will be reviewed as they arise.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 421 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
change in adiposity | baseline and 12 weeks
  measured by BMI, waist circumference, and body fat percentages (via Tanita scale)
change in blood pressure | baseline and 12 weeks
change in metabolic function | baseline and 12 weeks
  measured by fasting glucose, insulin and lipids

SECONDARY OUTCOMES:
change in dietary intake | basline and 12 weeks
  measured via screener, specifically fruits, vegetables, fiber
change in determinants of fruit and vegetable intake | basline and 12 weeks
  measured via LA Sprouts questionnaire (developed for this study), ie knowledge, preferences, self-efficacy, motivation

OTHER OUTCOMES:
change in school engagement | basline and 12 weeks
  measured via LA Sprouts questionnaire (developed for this study)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Spruijt-Metz, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Davis JN, Martinez LC, Spruijt-Metz D, Gatto NM. LA Sprouts: A 12-Week Gardening, Nutrition, and Cooking Randomized Control Trial Improves Determinants of Dietary Behaviors. J Nutr Educ Behav. 2016 Jan;48(1):2-11.e1. doi: 10.1016/j.jneb.2015.08.009. Epub 2015 Dec 10. PMID 26453367